CLINICAL TRIAL: NCT00424047
Title: The Official Title is A Multi-center, Randomized, Parallel-group, Double-blind, Placebo Controlled Study of CC-5013 Plus Dexamethasone Versus Dexamethasone Alone in Previously Treated Subjects With Multiple Myeloma.
Brief Title: A Study of CC-5013 Plus Dexamethasone Versus Dexamethasone Alone in Previously Treated Subjects With Multiple Myeloma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Celgene (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CC-5013-MM-010
Record Dates: First submitted 2007-01-17; First posted 2007-01-18 (Estimated); Results first posted 2015-03-04 (Estimated); Last update posted 2017-10-19 (Actual); Status verified 2017-09

CONDITIONS: Multiple Myeloma
Keywords: Multiple Myeloma; Celgene; Revlimid; CC-5013
MeSH Terms: conditions — Multiple Myeloma | interventions — Lenalidomide; Dexamethasone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- CC-5013 plus dexamethasone (Experimental): Arm A: Oral CC-5013 is initiated on Day 1 of Cycle 1 at a dose of 25 mg daily for 21 days every 28 days. Therefore, the subject will take a placebo identical in appearance to the CC-5013 capsule for week 4 of every 28 days. Oral pulse dexamethasone is administered at a dose of 40mg daily on Days 1-4, 9-12, and 17-20 of each 28 day cycle for Cycles 1 through 4. Beginning with Cycle 5, the oral dexamethasone dosing schedule will be reduced to 40mg daily for Days 1-4 every 28 days. In addition, oral CC-5013 placebo capsules will be administered for 28 days of every cycle.
  Interventions: Drug: CC-5013 plus dexamethasone
- Dexamethasone plus placebo (Experimental): Arm B: Oral pulse dexamethasone is administered at a dose of 40mg daily on Days 1-4, 9-12, and 17-20 of each 28 day cycle for Cycles 1 through 4. Beginning with Cycle 5, the oral dexamethasone dosing schedule will be reduced to 40mg daily for Days 1-4 every 28 days. In addition, oral placebo capsules will be administered for 28 days of every cycle.
  Interventions: Drug: Dexamethasone plus Placebo

INTERVENTIONS:
Drug: CC-5013 plus dexamethasone — 25 mg daily for 21 days every 28 days.
  Other Names: Revlimid; lenalidomide
  Arms: CC-5013 plus dexamethasone
Drug: Dexamethasone plus Placebo — Oral pulse dexamethasone is administered at a dose of 40mg daily on Days 1-4, 9-12, and 17-20 of each 28 day cycle for Cycles 1 through 4. Beginning with Cycle 5, the oral dexamethasone dosing schedule will be reduced to 40mg daily for Days 1-4 every 28 days. In addition, oral placebo capsules will be administered for 28 days of every cycle.
  Other Names: Dexamethasone; Placebo
  Arms: Dexamethasone plus placebo

SUMMARY:
To compare the efficacy of oral CC-5013 in combination with oral pulse high-dose dexamethasone to that of placebo and oral high-dose pulse dexamethasone as treatment for subjects with relapsed or refractory multiple myeloma."

ELIGIBILITY:
Inclusion Criteria:

* Prior or current diagnosis Durie-Salmon stage II or III multiple myeloma.
* Measurable levels of myeloma paraprotein in serum or urine (24-hour collection sample).
* Eastern Cooperative Oncology Group (ECOG) performance status score of 0,1, or 2
* Females of childbearing potential must have a negative serum or urine pregnancy test within 7 days of starting study drug

Exclusion Criteria:

* Prior development of disease progression during high-dose dexamethasone containing therapy
* Pregnant or lactating females
* The development of a desquamating rash while taking thalidomide
* Use of any standard/experimental anti-myeloma therapy within 28 days of randomization or use of any experimental non-drug therapy within 56 days of initiation of drug treatment
* Laboratory abnormalities: Absolute neutrophil count less than 1,000 cells/mm3
* Laboratory abnormalities: Platelet count < 75,000/mm3
* Laboratory abnormalities: Serum creatinine > 2.5 mg/dL
* Laboratory abnormalities: Serum Serum glutamic oxaloacetic transaminase (SGOT)/Aspartate aminotransferase (AST) or Serum glutamic pyruvic transaminase (SGPT)/Alanine aminotransferase (ALT) > 3.0 x upper limit of normal
* Laboratory abnormalities: Serum total bilirubin > 2.0 mg/dL
* Prior history of malignancies other than multiple myeloma unless the subject has been free of the disease for ≥ 3 years.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 351 (Actual)
Dates: Start 2003-01-01 (Actual); Primary Completion 2005-11-01 (Actual); Study Completion 2013-11-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Knight, MD, Study Director — Celgene Corporation
Locations (69):
- Australia (9):
  - Royal Prince Alfred Hospital, Camperdown, New South Wales
  - Peter MacCallum Cancer Centre Divsion of Haematology/Medical Oncology, East Melbourne, Victoria
  - The Alfred Hospital, Prahran, Victoria
  - Border Medical Oncology, Wodonga, Victoria
  - Box Hill Hospital, Box Hill
  - Frankston Hospital Oncology Research, Frankston
  - Royal Brisbane Hospital, Herston
  - The Royal Melbourne Hospital, Parkville
  - Mater Public Hospital, South Brisbane
- Austria (2):
  - University Hospital of Salzburg St Johanns Spital, Salzburg
  - Wilhelminenspital, Vienna
- Belgium (2):
  - CHU Saint-Luc, Brussels
  - UZ Gasthuisberg, Leuven
- France (7):
  - Centre Hospitalier Lyon Sud, Chemin Grand Revoyet
  - Hopital Claude Huriez, Lille
  - Centre Hospitalier Hotel-Dieu, Nantes
  - Hopital Saint-Loius, Paris
  - Chu de Bordeaux Groupe Hospitalier Sud, Pessac
  - CHU Purpan, Toulouse
  - CHU Nancy - Hopital Brabois, Vandœuvre-lès-Nancy
- Germany (9):
  - Universitaetsklinikum Charite, Berlin
  - Universitatsklinik ChariteMedizinische Fakultaet der HumboldtUniversitaet zu Berlin, Berlin
  - Universitaetsklinikum Dusseldorf Klinik fuer Haematologie, Düsseldorf
  - Universitaetsklinkum Erlangen, Erlangen
  - Klininkum der Johann-Wolfgang-Goethe-Universtat, Frankfurt am Main
  - Universitaetsklinikum Heidelberg Medizinische Klinik und Poliklinik V, Heidelberg
  - Klinikum der Univeristact Muenchen, München
  - Universitatsklinik Muenster Medizinische Klinik A, Münster
  - Universitaetsklinikum Tuebingen, Tübingen
- "Alexandras" General Hospital of Athens, Athens, Greece
- Ireland (4):
  - University Hospital GalwayHaematology Department, Galway, Co. Galway
  - Belfast City HospitalHaematology Department, Belfast
  - Hope Directorate Haematology Oncology Service St. James Hospital, Dublin
  - MidWestern Regional Hospital, Limerick
- Israel (4):
  - Rambam Medical Center, Haifa
  - Hadassah University Hospital, Jerusalem
  - Tel Aviv Sourasky Medical Center Department of Hematology, Tel Aviv
  - The Chaim Sheba Medical Center, Tel Litwinsky
- Italy (7):
  - Policlinico Sant'Orsola-Malpighi, Bologna
  - Azienda Ospedaliera San Martino, Genova
  - Ospedale Niguarda Ca Granda, Milan
  - Policlinico San Matteo, Pavia
  - Univerita La Sapien, Roma
  - Azienda Sanitaria Ospedaliera Molinette S. Giovanni Battista, Torio
  - Policlinico Universitario a Gesttione diretta di Udine, Udine
- Poland (3):
  - Institute of Internal Diseases University of Medicine, Gdansk
  - University School of Medicine, Lublin
  - Institute of Haematology and Blood Transfusion, Warsaw
- Spain (6):
  - Hospital Clinic, Barcelona
  - Hospital Universitario de la Princessa, Madrid
  - Hospital Doce de Octubre, Madrid
  - Clinica Universitaria de Navarra, Pamplona
  - Hospital Universitario de Salamanca, Salamanca
  - Hospital Universtario Marques de Valdecilla, Santander
- Sahlgrenska University Hospital Department of Hematology and Coagulation, Gothenburg, Sweden
- Switzerland (3):
  - Centre Hospitalier Universitaire Vaudois (CHUV), Lausanne
  - Kantonsspital St. Gallen, Sankt Gallen
  - Universitätsspital Zürich, Zurich
- Ukraine (8):
  - Cherkassy Regional Oncology Center, Cherkassy
  - Dnepropetrovsk City Clinical Hospital #4, Dnipro
  - Kiev Bone Marrow Transplantation Center Bone Marrow Department, Kiev
  - Institute of Hematology and Transfusiology of the UAMS Department of blood diseases, Kiev
  - Institute of Blood Pathology and Transfusion Medicine of the UAMS Hematology Department, Lviv
  - Institute of Blood Pathology and Transfusion Medicine of the UAMS, Lviv
  - Odess Regional Clinical Hospital, Odesa
  - Zhitomir Regional Clinical Hospital, Zhytomyr
- United Kingdom (3):
  - University College Hospital Trust, London, Bloomsbury
  - Bristol Haematology and Oncology Centre, Bristol
  - Haematology Dept, 4th Floor Thomas Guy House, London

REFERENCES:
- [Result] Dimopoulos M, Spencer A, Attal M, Prince HM, Harousseau JL, Dmoszynska A, San Miguel J, Hellmann A, Facon T, Foa R, Corso A, Masliak Z, Olesnyckyj M, Yu Z, Patin J, Zeldis JB, Knight RD; Multiple Myeloma (010) Study Investigators. Lenalidomide plus dexamethasone for relapsed or refractory multiple myeloma. N Engl J Med. 2007 Nov 22;357(21):2123-32. doi: 10.1056/NEJMoa070594. PMID 18032762
- [Derived] San-Miguel JF, Dimopoulos MA, Stadtmauer EA, Rajkumar SV, Siegel D, Bravo ML, Olesnyckyj M, Knight RD, Zeldis JB, Harousseau JL, Weber DM. Effects of lenalidomide and dexamethasone treatment duration on survival in patients with relapsed or refractory multiple myeloma treated with lenalidomide and dexamethasone. Clin Lymphoma Myeloma Leuk. 2011 Feb;11(1):38-43. doi: 10.3816/CLML.2010.n.120. PMID 21273172
- [Derived] Zangari M, Tricot G, Polavaram L, Zhan F, Finlayson A, Knight R, Fu T, Weber D, Dimopoulos MA, Niesvizky R, Fink L. Survival effect of venous thromboembolism in patients with multiple myeloma treated with lenalidomide and high-dose dexamethasone. J Clin Oncol. 2010 Jan 1;28(1):132-5. doi: 10.1200/JCO.2009.23.0169. Epub 2009 Nov 9. PMID 19901114
- [Derived] Wang M, Dimopoulos MA, Chen C, Cibeira MT, Attal M, Spencer A, Rajkumar SV, Yu Z, Olesnyckyj M, Zeldis JB, Knight RD, Weber DM. Lenalidomide plus dexamethasone is more effective than dexamethasone alone in patients with relapsed or refractory multiple myeloma regardless of prior thalidomide exposure. Blood. 2008 Dec 1;112(12):4445-51. doi: 10.1182/blood-2008-02-141614. Epub 2008 Sep 17. PMID 18799726
- See also: Link to CSR synopsis — http://www.celgene.com/research-development/clinical-trials/clinical-trials-data-sharing/clinical-study-report-csr-synopses/purposes-of-posting-clinical-study-report-csr-synopses

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 55 sites in Australia, Europe, and Israel. Eligible participants were randomized in a 1:1 ratio to: lenalidomide plus oral pulse high-dose dexamethasone or Placebo plus oral pulse high-dose dexamethasone.
Pre-assignment Details: A pre-specified interim analysis revealed a highly significant benefit favoring the lenalidomide/dexamethasone regimen, crossing the pre-specified O'Brien-Fleming superiority boundary. A decision was made to unblind the study allowing those receiving Placebo/dexamethasone to receive the lenalidomide/dexamethasone regimen.
Groups:
- Lenalidomide Plus Dexamethasone (Len/Dex): Lenalidomide 25 mg by mouth (PO) daily (QD) on Days 1 to 21 and a matching placebo capsule QD on Days 22 to 28 of each 28-day cycle.
  Pulse dexamethasone 40mg PO QD on Days 1-4, 9-12, and 17-20 of each 28-day cycle for cycles 1 through 4. Beginning with Cycle 5, dexamethasone dosing schedule was reduced to 40mg PO QD on Days 1 to 4 every 28 days for the remaining cycles.
- Placebo Plus Dexamethasone: Placebo PO daily on Days 1 to 28 of each 28 day cycle.
  Pulse dexamethasone 40mg PO QD on Days 1-4, 9-12, and 17-20 of each 28-day cycle for Cycles 1 through 4. Beginning with Cycle 5, dexamethasone dosing schedule was reduced to 40mg PO QD for Days 1-4 every 28 days.
  Participants with documented progressive disease were permitted to crossover to receive lenalidomide at the same doses mentioned.
  After the study was unblinded in August 2005 participants were given the option to add lenalidomide to their dexamethasone treatment regimen immediately or to add lenalidomide to their dexamethasone therapy at the time of disease progression.
Period: Blinded Treatment (Up to 03 Aug 2005)
Arm/Group | Lenalidomide Plus Dexamethasone (Len/Dex) | Placebo Plus Dexamethasone
Started | 176 | 175
Safety Population | 176 (Includes those who took at least one dose of study medication regimen) | 175 (Includes those who took at least one dose of study medication regimen)
Evaluable Population | 175 (1 participant excluded because they had no baseline M-protein assessment) | 171 (4 participants excluded because they had no baseline M-protein assessment)
Completed | 54 (54 participants ongoing and continuing on lenalidomide/dexamethasone treatment) | 19 (Ongoing and includes 15 participants who crossed over to lenalidomide/dexamethasone after unblinding)
Not Completed | 122 | 156
Not completed — Adverse Event | 18 | 12
Not completed — Progression of disease | 67 | 122
Not completed — Lack of therapeutic effect | 1 | 3
Not completed — Withdrawal by Subject | 23 | 8
Not completed — Death | 11 | 10
Not completed — Other | 2 | 1
Period: On Study at Time of Unblinding
Arm/Group | Lenalidomide Plus Dexamethasone (Len/Dex) | Placebo Plus Dexamethasone
Started | 176 (Refers to original treatment group assignment in the study.) | 175
Completed | 21 (Participants completed = those continuing on long term Lenalidomide and dexamethasone) | 8 (Participants completed = those continuing on long term dexamethasone)
Not Completed | 155 | 167
Not completed — Adverse Event | 22 | 12
Not completed — Progression of disease | 92 | 128
Not completed — Lack of Efficacy | 1 | 3
Not completed — Withdrawal by Subject | 24 | 9
Not completed — Death | 11 | 11
Not completed — Other | 5 | 4
Period: Long Term Extension (Up to 25 Jun 2013)
Arm/Group | Lenalidomide Plus Dexamethasone (Len/Dex) | Placebo Plus Dexamethasone
Started | 21 | 8 (2 participants opted to receive dex alone, 3 crossed over to Len/Dex and 3 added Len at a later date)
Completed | 0 | 0
Not Completed | 21 | 8
Not completed — Adverse Event | 1 | 0
Not completed — Death | 0 | 1
Not completed — Other | 12 | 4
Not completed — Progression of Disease | 7 | 3
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Population: Intent to treat population included all participants who were randomized
Groups:
- Lenalidomide Plus Dexamethasone: Lenalidomide 25 mg by mouth (PO) daily (QD) on Days 1 to 21 and a matching placebo capsule QD on Days 22 to 28 of each 28-day cycle.
  Dexamethasone 40mg PO QD on Days 1-4, 9-12, and 17-20 of each 28 day cycle for cycles 1 through 4. Beginning with Cycle 5, dexamethasone dosing schedule was reduced to 40mg PO QD on Days 1 to 4 every 28 days for the remaining cycles.
- Placebo Plus Dexamethasone: Placebo PO daily on Days 1 to 28 of each 28 day cycle.
  Dexamethasone 40mg PO QD on Days 1-4, 9-12, and 17-20 of each 28-day cycle for Cycles 1 through 4. Beginning with Cycle 5, dexamethasone dosing schedule was reduced to 40mg PO QD for Days 1-4 every 28 days.
- Total: Total of all reporting groups
Arm/Group | Lenalidomide Plus Dexamethasone | Placebo Plus Dexamethasone | Total
Number analyzed (Participants) | 176 | 175 | 351
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.2 (10.12) | 62.9 (8.80) | 62.6 (9.47)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 72 | 72 | 144
  Male | 104 | 103 | 207
Eastern Cooperative Oncology Group Performance Status [Number; unit: participants] — Eastern Cooperative Oncology Group (ECOG) Performance Status is used by doctors and researchers to assess how a participants' disease is progressing, assess how the disease affects the daily living activities of the participant and determine appropriate treatment and prognosis.
  participants
    0 = (Fully Active) | 78 | 65 | 143
    1 = (Restrictive but Ambulatory) | 72 | 79 | 151
    2 = Ambulatory unable to Work) | 23 | 27 | 50
    3 = (Limited Self-Care) | 0 | 1 | 1
    4 = (Completely Disabled) | 0 | 0 | 0
    Missing | 3 | 3 | 6
Number of Prior Anti-Myeloma Therapies [Number; unit: participants]
  1 Prior anti-myeloma therapy | 56 | 57 | 113
  2 or more prior anti-myeloma therapies | 120 | 118 | 238
Time from First Pathological Diagnosis [Median (Full Range); unit: years] | 3.4 [0.4 to 15.7] | 4.0 [0.3 to 26.6] | 3.7 [0.3 to 26.6]
Baseline multiple myeloma stage [Number; unit: participants] — The International Staging System divides myeloma into 3 stages based only on the serum beta-2 microglobulin and serum albumin levels.
  Stage I: Serum beta-2 microglobulin is less than 3.5 (mg/L) and the albumin level is above 3.5 (g/L);
  Stage II: Neither stage I or III, meaning that either:
  * The beta-2 microglobulin level is between 3.5 and 5.5 (with any albumin level), OR
  * The albumin is below 3.5 while the beta-2 microglobulin is less than 3.5
  Stage III: Serum beta-2 microglobulin is greater than 5.5.
  participants
    Stage I | 11 | 8 | 19
    Stage II | 50 | 57 | 107
    Stage III | 115 | 110 | 225

OUTCOME MEASURES:

1. Primary Outcome: Kaplan-Meier Estimate of Time to Tumor Progression (TTP)
Description: Time to progression was calculated as the time from randomization to the first occurrence of disease progression, as determined by a detailed review of all the myeloma response assessment data using the Bladé criteria (Bladé, 1998). Disease progression was also based on bone marrow findings, worsening lytic bone disease, progressively enlarging extramedullary plasmacytomas, or hypercalcemia.
Time Frame: From randomization up to cut-off date of 03 August 2005; up to 24 months
Population: Intent to treat included all participants who were randomized.
Measure: Median (95% Confidence Interval); unit: weeks
Groups:
- Lenalidomide Plus Dexamethasone: Lenalidomide 25 mg by mouth (PO) daily (QD) on Days 1 to 21 and a matching placebo capsule QD on Days 22 to 28 of each 28-day cycle.
  Pulse dexamethasone 40mg PO QD on Days 1-4, 9-12, and 17-20 of each 28 day cycle for cycles 1 through 4. Beginning with Cycle 5, dexamethasone dosing schedule was reduced to 40mg PO QD on Days 1 to 4 every 28 days for the remaining cycles.
- Placebo Plus Dexamethasone: Placebo PO daily on Days 1 to 28 of each 28 day cycle.
  Pulse dexamethasone 40mg PO QD on Days 1-4, 9-12, and 17-20 of each 28-day cycle for Cycles 1 through 4. Beginning with Cycle 5, dexamethasone dosing schedule was reduced to 40mg PO QD for Days 1-4 every 28 days.
Arm/Group | Lenalidomide Plus Dexamethasone | Placebo Plus Dexamethasone
Number analyzed (Participants) | 176 | 175
weeks | 52.1 [40.9 to NA] — Unable to provide as data not yet estimable | 20.1 [16.6 to 20.7]
Statistical Analysis 1: Comparison: Lenalidomide Plus Dexamethasone vs Placebo Plus Dexamethasone; Test type: Superiority or Other; p < 0.001, Log Rank; The p-value is based on an unstratified log rank test of survival curve differences between the treatment groups; Hazard Ratio (HR) = 0.324, 95% CI 2-sided [0.240 to 0.438] — Based on a proportional hazards model comparing the hazard functions associated with the treatment groups (Lenalidomide/Dex:Placebo/Dexamethasone)

2. Secondary Outcome: Kaplan-Meier Estimate of Overall Survival (OS)
Description: OS was calculated as the time from randomization to death from any cause. OS was censored at the last date that the participant was known to be alive for participants who were alive at the time of analysis and for participants who were lost to follow-up before death was documented.
Time Frame: Randomization to data cut off of 03 August 2005; up to 24 months
Population: Intent to Treat population includes all participants who were randomized.
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Lenalidomide Plus Dexamethasone | Placebo Plus Dexamethasone
Number analyzed (Participants) | 176 | 175
weeks | NA [NA to NA] — NA: Data not considered materialized or estimable at this time point | NA [71.6 to NA] — NA: Data not considered materialized or estimable at this time point
Statistical Analysis 1: Comparison: Lenalidomide Plus Dexamethasone vs Placebo Plus Dexamethasone; Test type: Superiority or Other; p = 0.105, Log Rank; The p-value is based on an unstratified log rank test of survival curve differences between the treatment groups; Hazard Ratio (HR) = 0.730, 95% CI 2-sided [0.498 to 1.070] — Based on a proportional hazards model comparing the hazard functions associated with the treatment groups (Lenalidomide/Dexamethasone:Placebo/Dexamethasone)

3. Secondary Outcome: Kaplan-Meier Estimate of Overall Survival (OS) (Later Cut-off Date of 02 March 2008)
Description: as for outcome 2
Time Frame: Randomization to data cut off of 02 March 2008; up to 51 months
Population: Intent to Treat population includes all participants who were randomized.
Measure: Median (95% Confidence Interval); unit: weeks
Groups:
- Placebo Plus Dexamethasone: Placebo PO daily on Days 1 to 28 of each 28 day cycle. Pulse dexamethasone 40 mg PO QD on Days 1-4, 9-12, and 17-20 of each 28-day cycle for Cycles 1 through 4. Beginning with Cycle 5, dexamethasone dosing schedule was reduced to 40 mg PO QD for Days 1-4 every 28 days.
  Participants with documented progressive disease were permitted to crossover to receive lenalidomide at the same doses mentioned.
  After the study was unblinded in August 2005 participants were given the option to add lenalidomide to their dexamethasone treatment regimen immediately or to add lenalidomide to their dexamethasone therapy at the time of disease progression.
Arm/Group | Lenalidomide Plus Dexamethasone | Placebo Plus Dexamethasone
Number analyzed (Participants) | 176 | 175
weeks | 161.9 [129.3 to 201.4] | 133.3 [101.6 to 174.0]
Statistical Analysis 1: Comparison: Lenalidomide Plus Dexamethasone vs Placebo Plus Dexamethasone; Test type: Superiority or Other; p = 0.302, Log Rank; The p-value is based on an unstratified log rank test of survival curve differences between the treatment groups; Hazard Ratio (HR) = 0.863, 95% CI 2-sided [0.651 to 1.143] — Based on a proportional hazards model comparing the hazard functions associated with the treatment groups (CC-5013/Dex:Placebo/Dex)

4. Secondary Outcome: Summary of Myeloma Response Rates Based on Best Response Assessment
Description: Complete Response (CR): Disappearance of monoclonal paraprotein and maintained for ≥ 6 weeks . Remission Response (RR):75-99% reduction in the level of the serum monoclonal paraprotein compared to baseline; 90-99% reduction in 24-hr urinary light chain excretion. Partial Response (PR): 50-74% reduction in the level of monoclonal paraprotein compared to baseline; 50-89% reduction in 24-hr urinary light chain excretion. Stable Disease (SD): Criteria for PR or PD have not been met. Plateau Phase: If PR, stable monoclonal paraprotein values (within 25% above or below nadir)/stable soft tissue plasmacytomas maintained for at least 3 months. Progressive Disease (PD): Reappearance of serum or urinary monoclonal paraprotein on immunofixation or electrophoresis on two consecutive occasions at least one week apart. Increase of percentage of plasma cells in bone marrow aspirate or biopsy to ≥ 5%. Development of at least one new lytic bone lesion or soft tissue plasmacytoma.
Time Frame: Randomization to 03 August 2005; up to 24 months
Population: Intent to Treat Population includes all participants who were randomized
Measure: Number; unit: percentage of participants
Arm/Group | Lenalidomide Plus Dexamethasone | Placebo Plus Dexamethasone
Number analyzed (Participants) | 176 | 175
percentage of participants
  Complete Response (CR) | 15.3 | 4.0
  Partial Response (PR) | 43.8 | 19.4
  Stable Disease (SD) | 29.0 | 56.6
  Progressive Disease (PD) | 2.8 | 14.3
  Not Evaluable (NE) those without response data | 9.1 | 5.7
Statistical Analysis 1: Comparison: Lenalidomide Plus Dexamethasone vs Placebo Plus Dexamethasone; Test type: Superiority or Other; p < 0.001, Wilcoxon (Mann-Whitney); Probability from Wilcoxon rank sum test

5. Secondary Outcome: Myeloma Response Rates Based on the Reviewers Best Response Assessment (Later Cut-off Date of 02 March 2008)
Description: as for outcome 4
Time Frame: Randomization to data cut-off of 02 Mar 2008; up to 51 months
Population: Intent to Treat Population includes all participants who were randomized
Measure: Number; unit: percentage of participants
Arm/Group | Lenalidomide Plus Dexamethasone | Placebo Plus Dexamethasone
Number analyzed (Participants) | 176 | 175
percentage of participants
  Complete Response (CR) | 17.0 | 4.0
  Partial Response (PR) | 42.6 | 19.4
  Stable Disease (SD) | 28.4 | 56.6
  Progressive Disease (PD) | 3.4 | 14.3
  Not Evaluable (NE) those without response data | 8.5 | 5.7
Statistical Analysis 1: Comparison: Lenalidomide Plus Dexamethasone vs Placebo Plus Dexamethasone; Test type: Superiority or Other; p < 0.001, Wilcoxon (Mann-Whitney); Probability from Wilcoxon rank sum test

6. Secondary Outcome: Number of Participants With Adverse Events (AE)
Description: An AE is any sign, symptom, illness, or diagnosis that appears or worsens during the course of the study. Treatment-emergent AEs (TEAEs) are any AE occurring or worsening on or after the first treatment of the study drug and within 30 days after the last cycle end date of study drug. A serious AE = any AE which results in death; is life-threatening; requires or prolongs existing inpatient hospitalization; results in persistent or significant disability is a congenital anomaly/birth defect; constitutes an important medical event.
  The severity of AEs were graded according to the National Cancer Institute (NCI) Common Terminology Criteria for AEs (CTCAE, Version 2.0): Grade 1 = Mild (no limitation in activity or intervention required); Grade 2 = Moderate (some limitation in activity; no/minimal medical intervention required); Grade 3 = Severe (marked limitation in activity; medical intervention required, hospitalization possible); Grade 4 = Life-threatening; Grade 5 = Death.
Time Frame: From first dose of study drug through to 30 days after the last dose, until the data cut-off date of 25 June 2013; up to 90 months
Population: The safety population includes all participants who received at least one dose of study drug regimen
Measure: Number; unit: participants
Arm/Group | Lenalidomide Plus Dexamethasone | Placebo Plus Dexamethasone
Number analyzed (Participants) | 176 | 175
participants
  ≥ 1 Adverse Event | 176 | 175
  ≥ 1 Serious Adverse Event | 105 | 79
  ≥ 1 AE leading to study drug discontinuation | 46 | 31
  ≥ 1 AE leading to dose reduction or interruption | 137 | 100
  ≥ 1 Drug-Related Adverse Event | 160 | 151
  ≥ 1 Drug-Related Serious Adverse Event | 54 | 30
  ≥Death within ≤ 30 days of last dose of study drug | 17 | 20
  ≥ 1 Grade 1 or Higher Adverse Event | 176 | 175
  ≥ 1 Grade 2 or Higher Adverse Event | 168 | 167
  ≥ 1 Grade 3 or Higher Adverse Event | 146 | 119
  ≥ 1 Grade 4 or Higher Adverse Event | 52 | 37

7. Secondary Outcome: Time to First Symptomatic Skeletal-related Event (SRE) (Clinical Need for Radiation or Surgery to Bone)
Description: Time from randomization to the date of the first occurrence of a symptomatic SRE (clinical need for radiotherapy or surgery to bone).
Time Frame: Up to unblinding data cut off of 03 August 2005; up to 24 months
Population: Analysis not performed due to an insufficient number of participants with SRE
Measure: Number; unit: participants
Arm/Group | Lenalidomide Plus Dexamethasone | Placebo Plus Dexamethasone
Number analyzed (Participants) | 176 | 175
participants | NA — There were an insufficient number of participants with SRE events and no analysis was conducted. | NA — There were an insufficient number of participants with SRE events and no analysis was conducted.

8. Post Hoc Outcome: Kaplan-Meier Estimate of Duration of Response
Description: Duration of response was calculated for responders and defined as the time from the first observation of a response (e.g., the first time that the appropriate decrease in M-protein level was observed for confirmed responders) to the first documented progression or relapse. Response duration was censored at the last adequate assessment showing evidence of no progression.
Time Frame: Up to data cut off of 03 August 2005; up to 24 months
Population: Intent to Treat population includes all participants who were randomized to study drug.
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Lenalidomide Plus Dexamethasone | Placebo Plus Dexamethasone
Number analyzed (Participants) | 104 | 41
weeks | 67.6 [42.1 to NA] — NA: Data not considered materialized or estimable at this time point | 33.3 [22.1 to 51.6]
Statistical Analysis 1: Comparison: Lenalidomide Plus Dexamethasone vs Placebo Plus Dexamethasone; Test type: Superiority or Other; p = 0.021, Log Rank; The p-value is based on an unstratified log rank test of survival curve differences between the treatment groups; Hazard Ratio (HR) = 0.558, 95% CI 2-sided [0.338 to 0.921] — Based on a proportional hazards model comparing the hazard functions associated with the treatment groups (lenalidomide/dexamethasone : placebo/dexamethasone)

9. Primary Outcome: Kaplan-Meier Estimate of Time to Tumor Progression (TTP) (Later Cut-off Date of 02 Mar 2008)
Description: as for outcome 1
Time Frame: From randomization up to cut-off date of 02 March 2008; up to 51 months
Population: Intent to treat included all participants who were randomized.
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Lenalidomide Plus Dexamethasone | Placebo Plus Dexamethasone
Number analyzed (Participants) | 176 | 175
weeks | 52.4 [40.9 to 85.6] | 20.1 [16.6 to 20.7]
Statistical Analysis 1: Comparison: Lenalidomide Plus Dexamethasone vs Placebo Plus Dexamethasone; Test type: Superiority or Other; p < 0.001, Log Rank — The p-value is based on an unstratified log rank test of survival curve differences between the treatment groups; Hazard Ratio (HR) = 0.362, 95% CI 2-sided [0.27 to 0.478] — [estimate comment as in outcome 3, analysis 1]

10. Secondary Outcome: Time to First Worsening on the Eastern Cooperative Oncology Group (ECOG) Performance Scale
Description: The time to first worsening of the ECOG performance status was calculated as the time from randomization to the date of the first worsening compared with the last ECOG evaluation obtained prior to randomization. Data were censored at the last date that the participant was known to be unchanged or improved from before randomization for the participants who had not had worsened at the time of the analysis and for the patients who were lost to follow-up before worsening in the ECOG performance status was documented.
Time Frame: Randomization to cut off date of 03 August 2005; up to 24 months
Population: Intent to Treat includes all participants who were randomized to study drug; a total of six ECOG scores were missing at the time of the Aug 2005 cut-off.
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Lenalidomide Plus Dexamethasone | Placebo Plus Dexamethasone
Number analyzed (Participants) | 173 | 172
weeks | 10.1 [8.1 to 16.1] | 12.3 [10.1 to 24.1]
Statistical Analysis 1: Comparison: Lenalidomide Plus Dexamethasone vs Placebo Plus Dexamethasone; Test type: Superiority or Other; p = 0.271, Log Rank — The p-value is based on an unstratified log rank test of survival curve differences between the treatment groups; Hazard Ratio (HR) = 1.166, 95% CI 2-sided [0.887 to 1.532] — Based on a proportional hazards model comparing the hazard functions associated with the treatment groups (lenalidomide/dexamethasone: placebo/dexamethasone)

11. Secondary Outcome: Time to First Worsening on the Eastern Cooperative Oncology Group (ECOG) Performance Scale (Later Cut-off Date of 02 March 2008)
Description: as for outcome 10
Time Frame: Randomization to cut off date of 02 March 2008; up to 51 months
Population: Intent to Treat includes all participants who were randomized to study drug; six ECOG scores were missing at the March 2008 cut-off.
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Lenalidomide Plus Dexamethasone | Placebo Plus Dexamethasone
Number analyzed (Participants) | 173 | 172
weeks | 10.1 [8.1 to 16.1] | 12.3 [10.1 to 24.1]
Statistical Analysis 1: Comparison: Lenalidomide Plus Dexamethasone vs Placebo Plus Dexamethasone; Test type: Superiority or Other; p = 0.359, Log Rank — The p-value is based on an unstratified log rank test of survival curve differences between the treatment groups; Hazard Ratio (HR) = 1.135, 95% CI 2-sided [0.866 to 1.486] — [estimate comment as in outcome 3, analysis 1]

12. Post Hoc Outcome: Kaplan-Meier Estimate of Duration of Response (Cut-off at a Later Date of 03 March 2008)
Description: as for outcome 8
Time Frame: Up to data cut off of 03 Mar 2008; up to 51 months
Population: Intent to Treat population includes all participants who were randomized to study drug.
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Lenalidomide Plus Dexamethasone | Placebo Plus Dexamethasone
Number analyzed (Participants) | 105 | 41
weeks | 68.1 [42.1 to 105.6] | 33.3 [22.1 to 51.6]
Statistical Analysis 1: Comparison: Lenalidomide Plus Dexamethasone vs Placebo Plus Dexamethasone; Test type: Superiority or Other; p = 0.032, Log Rank; The p-value is based on an unstratified log rank test of survival curve differences between the treatment groups; Hazard Ratio (HR) = 0.619, 95% CI 2-sided [0.398 to 0.964] — [estimate comment as in outcome 3, analysis 1]

ADVERSE EVENTS:
Time Frame: From first dose of study drug to 30 days after the last visit. Up to 25 Jun 2013 (90 Months).
Description: Includes adverse events for those who received Lenalidomide after unblinding.
Arm/Group | Lenalidomide Plus Dexamethasone | Placebo Plus Dexamethasone
Serious Adverse Events (participants affected / at risk) | 105/176 | 79/175
Other Adverse Events (participants affected / at risk) | 175/176 | 173/175
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Lenalidomide Plus Dexamethasone (N=176) | Placebo Plus Dexamethasone (N=175)
PNEUMONIA NOS (Infections and infestations) | 11 | 7
RESPIRATORY TRACT INFECTION NOS (Infections and infestations) | 4 | 7
SEPSIS NOS (Infections and infestations) | 3 | 3
SEPTIC SHOCK (Infections and infestations) | 2 | 2
UPPER RESPIRATORY TRACT INFECTION NOS (Infections and infestations) | 4 | 0
BRONCHOPNEUMONIA NOS (Infections and infestations) | 3 | 0
CELLULITIS (Infections and infestations) | 1 | 2
ARTHRITIS BACTERIAL (Infections and infestations) | 2 | 0
BRONCHITIS ACUTE NOS (Infections and infestations) | 2 | 0
HERPES ZOSTER (Infections and infestations) | 2 | 0
HERPES ZOSTER OPHTHALMIC (Infections and infestations) | 1 | 1
LOBAR PNEUMONIA NOS (Infections and infestations) | 2 | 0
PNEUMOCYSTIS CARINII PNEUMONIA (Infections and infestations) | 2 | 0
PNEUMONIA PNEUMOCOCCAL (Infections and infestations) | 1 | 1
URINARY TRACT INFECTION NOS (Infections and infestations) | 1 | 1
UROSEPSIS (Infections and infestations) | 1 | 1
BACTERAEMIA (Infections and infestations) | 0 | 1
BACTERIAL SEPSIS (Infections and infestations) | 1 | 0
BRONCHITIS CHRONIC NOS (Infections and infestations) | 0 | 1
BURSITIS INFECTIVE NOS (Infections and infestations) | 1 | 0
CENTRAL LINE INFECTION (Infections and infestations) | 1 | 0
CLOSTRIDIUM DIFFICILE SEPSIS (Infections and infestations) | 1 | 0
ESCHERICHIA URINARY TRACT INFECTION (Infections and infestations) | 0 | 1
GASTROINTESTINAL INFECTION NOS (Infections and infestations) | 0 | 1
LOWER RESPIRATORY TRACT INFECTION NOS (Infections and infestations) | 1 | 0
LUNG INFECTION NOS (Infections and infestations) | 0 | 1
MENINGITIS (Infections and infestations) | 1 | 0
MENINGITIS PNEUMOCOCCAL (Infections and infestations) | 1 | 0
NECROTISING FASCIITIS NOS (Infections and infestations) | 1 | 0
OTITIS MEDIA NOS (Infections and infestations) | 1 | 0
PNEUMONIA BACTERIAL NOS (Infections and infestations) | 1 | 0
PNEUMONIA LEGIONELLA (Infections and infestations) | 1 | 0
PYELONEPHRITIS ACUTE NOS (Infections and infestations) | 1 | 0
RESPIRATORY TRACT INFECTION VIRAL NOS (Infections and infestations) | 1 | 0
SALMONELLA INFECTION NOS (Infections and infestations) | 1 | 0
SINUSITIS NOS (Infections and infestations) | 1 | 0
STAPHYLOCOCCAL INFECTION (Infections and infestations) | 1 | 0
STAPHYLOCOCCAL SEPSIS (Infections and infestations) | 0 | 1
STREPTOCOCCAL SEPSIS (Infections and infestations) | 1 | 1
URINARY TRACT INFECTION BACTERIAL (Infections and infestations) | 1 | 0
PYREXIA (General disorders) | 6 | 7
GENERAL PHYSICAL HEALTH DETERIORATION (General disorders) | 4 | 1
ASTHENIA (General disorders) | 2 | 1
DIFFICULTY IN WALKING (General disorders) | 2 | 0
MULTI-ORGAN FAILURE (General disorders) | 2 | 0
OEDEMA PERIPHERAL (General disorders) | 2 | 0
PERFORMANCE STATUS DECREASED (General disorders) | 1 | 1
CATHETER SITE INFLAMMATION (General disorders) | 1 | 0
GRANULOMA NOS (General disorders) | 1 | 0
INFLUENZA LIKE ILLNESS (General disorders) | 0 | 1
NECROSIS NOS (General disorders) | 0 | 1
PAIN NOS (General disorders) | 0 | 1
SUDDEN DEATH (General disorders) | 1 | 0
BACK PAIN (Musculoskeletal and connective tissue disorders) | 5 | 1
BONE PAIN (Musculoskeletal and connective tissue disorders) | 5 | 0
MUSCLE WEAKNESS NOS (Musculoskeletal and connective tissue disorders) | 1 | 3
OSTEONECROSIS (Musculoskeletal and connective tissue disorders) | 3 | 1
PATHOLOGICAL FRACTURE (Musculoskeletal and connective tissue disorders) | 1 | 2
PAIN IN LIMB (Musculoskeletal and connective tissue disorders) | 1 | 1
CHEST WALL PAIN (Musculoskeletal and connective tissue disorders) | 1 | 0
JOINT SWELLING (Musculoskeletal and connective tissue disorders) | 1 | 0
MYALGIA (Musculoskeletal and connective tissue disorders) | 1 | 0
MYOPATHY (Musculoskeletal and connective tissue disorders) | 0 | 1
MYOPATHY STEROID (Musculoskeletal and connective tissue disorders) | 1 | 0
OSTEOPOROSIS NOS (Musculoskeletal and connective tissue disorders) | 0 | 1
PAIN IN JAW (Musculoskeletal and connective tissue disorders) | 1 | 0
SPONDYLITIS NOS (Musculoskeletal and connective tissue disorders) | 1 | 0
DEEP VEIN THROMBOSIS (Vascular disorders) | 8 | 6
HYPOTENSION NOS (Vascular disorders) | 2 | 2
PHLEBITIS NOS (Vascular disorders) | 1 | 2
VENOUS THROMBOSIS NOS LIMB (Vascular disorders) | 2 | 1
PERIPHERAL ISCHAEMIA (Vascular disorders) | 2 | 0
CIRCULATORY COLLAPSE (Vascular disorders) | 1 | 0
PHLEBITIS SUPERFICIAL (Vascular disorders) | 1 | 0
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 7 | 2
ACUTE RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 1 | 1
BRONCHITIS NOS (Respiratory, thoracic and mediastinal disorders) | 1 | 1
BRONCHOSPASM NOS (Respiratory, thoracic and mediastinal disorders) | 1 | 1
RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 2 | 0
ACUTE RESPIRATORY DISTRESS SYNDROME (Respiratory, thoracic and mediastinal disorders) | 1 | 0
BRONCHOPNEUMOPATHY (Respiratory, thoracic and mediastinal disorders) | 0 | 1
COUGH (Respiratory, thoracic and mediastinal disorders) | 1 | 0
DYSPNOEA NOS (Respiratory, thoracic and mediastinal disorders) | 0 | 1
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 0 | 1
LUNG CONSOLIDATION (Respiratory, thoracic and mediastinal disorders) | 1 | 0
MAXILLARY SINUSITIS (Respiratory, thoracic and mediastinal disorders) | 0 | 1
PNEUMONIA ASPIRATION (Respiratory, thoracic and mediastinal disorders) | 0 | 1
PULMONARY CONGESTION (Respiratory, thoracic and mediastinal disorders) | 1 | 0
DIARRHOEA NOS (Gastrointestinal disorders) | 2 | 2
CONSTIPATION (Gastrointestinal disorders) | 1 | 1
MELAENA (Gastrointestinal disorders) | 0 | 2
OESOPHAGEAL VARICES HAEMORRHAGE (Gastrointestinal disorders) | 1 | 1
OESOPHAGITIS NOS (Gastrointestinal disorders) | 1 | 1
UPPER GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 0 | 2
ABDOMINAL PAIN NOS (Gastrointestinal disorders) | 1 | 0
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 0 | 1
CAECITIS (Gastrointestinal disorders) | 1 | 0
COLOVESICAL FISTULA (Gastrointestinal disorders) | 0 | 1
DIVERTICULITIS INTESTINAL (Gastrointestinal disorders) | 0 | 1
DIVERTICULITIS NOS (Gastrointestinal disorders) | 1 | 0
GASTRIC ULCER (Gastrointestinal disorders) | 0 | 1
GASTRITIS NOS (Gastrointestinal disorders) | 1 | 0
GASTROENTERITIS NOS (Gastrointestinal disorders) | 1 | 0
GASTROINTESTINAL HAEMORRHAGE NOS (Gastrointestinal disorders) | 1 | 0
NAUSEA (Gastrointestinal disorders) | 1 | 0
OESOPHAGITIS ULCERATIVE (Gastrointestinal disorders) | 0 | 1
PEPTIC ULCER HAEMORRHAGE (Gastrointestinal disorders) | 1 | 0
VOMITING NOS (Gastrointestinal disorders) | 1 | 0
CEREBROVASCULAR ACCIDENT (Nervous system disorders) | 3 | 2
MEMORY IMPAIRMENT (Nervous system disorders) | 1 | 1
SPINAL CORD COMPRESSION NOS (Nervous system disorders) | 2 | 0
ATAXIA (Nervous system disorders) | 1 | 0
BRAIN OEDEMA (Nervous system disorders) | 0 | 1
CEREBRAL ISCHAEMIA (Nervous system disorders) | 1 | 0
ENCEPHALITIS NOS (Nervous system disorders) | 0 | 1
EPIDURITIS (Nervous system disorders) | 0 | 1
HYPOAESTHESIA (Nervous system disorders) | 0 | 1
INTRACRANIAL PRESSURE INCREASED NOS (Nervous system disorders) | 0 | 1
LEUKOENCEPHALOPATHY (Nervous system disorders) | 1 | 0
PERIPHERAL MOTOR NEUROPATHY (Nervous system disorders) | 0 | 1
PERIPHERAL NEUROPATHY NOS (Nervous system disorders) | 1 | 0
POLYNEUROPATHY NOS (Nervous system disorders) | 1 | 0
SUBDURAL HAEMATOMA (Nervous system disorders) | 0 | 1
TREMOR (Nervous system disorders) | 0 | 1
ANAEMIA NOS (Blood and lymphatic system disorders) | 4 | 1
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 2 | 3
NEUTROPENIA (Blood and lymphatic system disorders) | 3 | 1
FEBRILE NEUTROPENIA (Blood and lymphatic system disorders) | 4 | 0
PANCYTOPENIA (Blood and lymphatic system disorders) | 0 | 2
HYPERVISCOSITY SYNDROME (Blood and lymphatic system disorders) | 1 | 0
THROMBOTIC THROMBOCYTOPENIC PURPURA (Blood and lymphatic system disorders) | 1 | 0
RENAL FAILURE ACUTE (Renal and urinary disorders) | 4 | 3
RENAL FAILURE NOS (Renal and urinary disorders) | 3 | 4
RENAL IMPAIRMENT NOS (Renal and urinary disorders) | 0 | 2
FANCONI SYNDROME ACQUIRED (Renal and urinary disorders) | 1 | 0
OLIGURIA (Renal and urinary disorders) | 0 | 1
RENAL COLIC (Renal and urinary disorders) | 1 | 0
RENAL FAILURE ACUTE ON CHRONIC (Renal and urinary disorders) | 1 | 0
URINARY RETENTION (Renal and urinary disorders) | 1 | 0
PULMONARY OEDEMA NOS (Cardiac disorders) | 1 | 3
ATRIAL FIBRILLATION (Cardiac disorders) | 2 | 1
MYOCARDIAL INFARCTION (Cardiac disorders) | 1 | 2
ACUTE CORONARY SYNDROME (Cardiac disorders) | 1 | 0
ACUTE MYOCARDIAL INFARCTION (Cardiac disorders) | 1 | 0
ANGINA UNSTABLE (Cardiac disorders) | 0 | 1
CARDIAC FAILURE ACUTE (Cardiac disorders) | 0 | 1
CARDIAC FAILURE CONGESTIVE (Cardiac disorders) | 1 | 0
CARDIAC FAILURE NOS (Cardiac disorders) | 0 | 1
CARDIO-RESPIRATORY ARREST (Cardiac disorders) | 0 | 1
CORONARY ARTERY STENOSIS (Cardiac disorders) | 0 | 1
MYOCARDIAL ISCHAEMIA (Cardiac disorders) | 0 | 1
VENTRICULAR BIGEMINY (Cardiac disorders) | 0 | 1
HYPERGLYCAEMIA NOS (Metabolism and nutrition disorders) | 3 | 2
DEHYDRATION (Metabolism and nutrition disorders) | 1 | 1
ELECTROLYTE IMBALANCE (Metabolism and nutrition disorders) | 2 | 0
HYPERCALCAEMIA (Metabolism and nutrition disorders) | 0 | 3
HYPOCALCAEMIA (Metabolism and nutrition disorders) | 1 | 1
DIABETES MELLITUS INADEQUATE CONTROL (Metabolism and nutrition disorders) | 1 | 0
DIABETES MELLITUS NOS (Metabolism and nutrition disorders) | 0 | 1
DEPRESSION (Psychiatric disorders) | 3 | 1
CONFUSIONAL STATE (Psychiatric disorders) | 1 | 1
BIPOLAR DISORDER (Psychiatric disorders) | 0 | 1
DELIRIUM (Psychiatric disorders) | 0 | 1
INSOMNIA (Psychiatric disorders) | 1 | 0
MANIA (Psychiatric disorders) | 0 | 1
MENTAL DISORDER NOS (Psychiatric disorders) | 0 | 1
BASAL CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
BREAST CANCER IN SITU (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
GLIOBLASTOMA MULTIFORME (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
LUNG ADENOCARCINOMA NOS (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
NEOPLASM NOS (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
PROSTATE CANCER NOS (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
TRANSITIONAL CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
FEMUR FRACTURE (Injury, poisoning and procedural complications) | 2 | 0
JOINT DISLOCATION (Injury, poisoning and procedural complications) | 1 | 0
POST PROCEDURAL COMPLICATION (Injury, poisoning and procedural complications) | 1 | 0
POST PROCEDURAL PAIN (Injury, poisoning and procedural complications) | 1 | 0
SPINAL FRACTURE NOS (Injury, poisoning and procedural complications) | 0 | 1
THORACIC VERTEBRAL FRACTURE (Injury, poisoning and procedural complications) | 0 | 1
BLOOD CREATININE INCREASED (Investigations) | 0 | 1
BODY TEMPERATURE INCREASED (Investigations) | 0 | 1
C-REACTIVE PROTEIN INCREASED (Investigations) | 0 | 1
INTERNATIONAL NORMALISED RATIO DECREASED (Investigations) | 1 | 0
WEIGHT DECREASED (Investigations) | 1 | 0
CHOLELITHIASIS (Hepatobiliary disorders) | 2 | 0
CHOLECYSTITIS ACUTE NOS (Hepatobiliary disorders) | 1 | 0
HEPATIC FAILURE (Hepatobiliary disorders) | 1 | 0
ACQUIRED HYPOTHYROIDISM (Endocrine disorders) | 0 | 1
ADRENAL INSUFFICIENCY NOS (Endocrine disorders) | 0 | 1
CORNEAL ULCER (Eye disorders) | 1 | 0
EXOPHTHALMOS NOS (Eye disorders) | 0 | 1
BREAST MICROCALCIFICATION (Reproductive system and breast disorders) | 1 | 0
LUNG SQUAMOUS CELL CARCINOMA, STAGE UNSPECIFIED (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
LEUKOPLAKIA NOS (Skin and subcutaneous tissue disorders) | 1 | 0
PHLEBOTHROMBOSIS (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Lenalidomide Plus Dexamethasone (N=176) | Placebo Plus Dexamethasone (N=175)
NEUTROPENIA (Blood and lymphatic system disorders) | 71 | 17
ANAEMIA (Blood and lymphatic system disorders) | 52 | 49
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 33 | 19
LEUKOPENIA (Blood and lymphatic system disorders) | 21 | 11
LYMPHOPENIA (Blood and lymphatic system disorders) | 17 | 9
VERTIGO (Ear and labyrinth disorders) | 12 | 8
CUSHINGOID (Endocrine disorders) | 9 | 4
VISION BLURRED (Eye disorders) | 13 | 13
CONSTIPATION (Gastrointestinal disorders) | 71 | 41
DIARRHOEA NOS (Gastrointestinal disorders) | 67 | 45
NAUSEA (Gastrointestinal disorders) | 40 | 20
DYSPEPSIA (Gastrointestinal disorders) | 23 | 23
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 22 | 11
VOMITING NOS (Gastrointestinal disorders) | 20 | 12
ABDOMINAL PAIN NO (Gastrointestinal disorders) | 16 | 10
STOMATITIS (Gastrointestinal disorders) | 11 | 6
DRY MOUTH (Gastrointestinal disorders) | 10 | 5
GASTRITIS NOS (Gastrointestinal disorders) | 9 | 4
GASTROENTERITIS NOS (Gastrointestinal disorders) | 9 | 5
ASTHENIA (General disorders) | 64 | 46
FATIGUE (General disorders) | 51 | 41
PYREXIA (General disorders) | 50 | 40
OEDEMA PERIPHERAL (General disorders) | 42 | 34
OEDEMA NOS (General disorders) | 22 | 15
LETHARGY (General disorders) | 15 | 4
CHEST PAIN (General disorders) | 11 | 7
UPPER RESPIRATORY TRACT INFECTION NOS (Infections and infestations) | 29 | 16
URINARY TRACT INFECTION NOS (Infections and infestations) | 15 | 13
INFLUENZA (Infections and infestations) | 10 | 8
ORAL CANDIDIASIS (Infections and infestations) | 10 | 9
LOWER RESPIRATORY TRACT INFECTION NOS (Infections and infestations) | 9 | 11
RESPIRATORY TRACT INFECTION NOS (Infections and infestations) | 9 | 6
HERPES SIMPLEX (Infections and infestations) | 8 | 12
SINUSITIS NOS (Infections and infestations) | 6 | 9
WEIGHT DECREASED (Investigations) | 49 | 46
WEIGHT INCREASED (Investigations) | 17 | 24
ANOREXIA (Metabolism and nutrition disorders) | 25 | 14
HYPOKALAEMIA (Metabolism and nutrition disorders) | 20 | 10
HYPERGLYCAEMIA NOS (Metabolism and nutrition disorders) | 19 | 22
HYPOCALCAEMIA (Metabolism and nutrition disorders) | 16 | 5
HYPOPHOSPHATAEMIA (Metabolism and nutrition disorders) | 11 | 2
HYPERURICAEMIA (Metabolism and nutrition disorders) | 4 | 10
MUSCLE CRAMP (Musculoskeletal and connective tissue disorders) | 56 | 36
BACK PAIN (Musculoskeletal and connective tissue disorders) | 45 | 29
BONE PAIN (Musculoskeletal and connective tissue disorders) | 34 | 24
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 33 | 28
MUSCLE WEAKNESS NOS (Musculoskeletal and connective tissue disorders) | 30 | 28
PAIN IN LIMB (Musculoskeletal and connective tissue disorders) | 27 | 20
MYALGIA (Musculoskeletal and connective tissue disorders) | 18 | 16
CHEST WALL PAIN (Musculoskeletal and connective tissue disorders) | 11 | 14
HEADACHE (Nervous system disorders) | 41 | 35
TREMOR (Nervous system disorders) | 39 | 14
DIZZINESS (Nervous system disorders) | 36 | 16
PARAESTHESIA (Nervous system disorders) | 29 | 29
DYSGEUSIA (Nervous system disorders) | 20 | 16
HYPOAESTHESIA (Nervous system disorders) | 15 | 7
SOMNOLENCE (Nervous system disorders) | 8 | 10
INSOMNIA (Psychiatric disorders) | 51 | 63
DEPRESSION (Psychiatric disorders) | 19 | 18
CONFUSIONAL STATE (Psychiatric disorders) | 14 | 10
ANXIETY (Psychiatric disorders) | 11 | 14
MOOD ALTERATION NOS (Psychiatric disorders) | 5 | 10
COUGH (Respiratory, thoracic and mediastinal disorders) | 41 | 41
DYSPNOEA NOS (Respiratory, thoracic and mediastinal disorders) | 36 | 22
NASOPHARYNGITIS (Respiratory, thoracic and mediastinal disorders) | 35 | 23
BRONCHITIS NOS (Respiratory, thoracic and mediastinal disorders) | 27 | 26
PHARYNGITIS (Respiratory, thoracic and mediastinal disorders) | 27 | 16
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 12 | 17
HICCUPS (Respiratory, thoracic and mediastinal disorders) | 10 | 8
RHINITIS NOS (Respiratory, thoracic and mediastinal disorders) | 5 | 9
RASH NOS (Skin and subcutaneous tissue disorders) | 24 | 9
SWEATING INCREASED (Skin and subcutaneous tissue disorders) | 17 | 16
DRY SKIN (Skin and subcutaneous tissue disorders) | 16 | 6
PRURITUS (Skin and subcutaneous tissue disorders) | 11 | 9
ERYTHEMA (Skin and subcutaneous tissue disorders) | 8 | 13
HYPERTENSION NOS (Vascular disorders) | 17 | 11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Investigator has the right to publish and/or present study data after multicentric publication or one year has elapsed until completion of this multicentric study provided that he/she (i) furnishes the sponsor a copy of any proposed publication or presentation before its submission, (ii) deletes any sponsor's confidential data as pointed out by sponsor, and (iii) delays any submission for generally up to ninety (90) days to permit the preparation and filing of intellectual property applications.